CLINICAL TRIAL: NCT00951912
Title: The Study of the Effects of Soy Isoflavones on the Metabolism of Glucose and Lipids in Postmenopausal Chinese Women With Impaired Glucose Regulation
Brief Title: The Effects of Soy Isoflavones to Improve the Metabolism of Glucose and Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese Nutrition Society (Unknown); Danone Institute International (Other); Department of Health of Guangdong Province (Unknown)
Responsible Party: Principal Investigator, yanbinye, Associate professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: yanbinye
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: genistein; daidzein; impaired glucose regulation; glucose metabolism; lipids metabolism; inflammation; women
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — daidzein; Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 10g soy protein isolated powder patch by mouth everyday for 6months
  Interventions: Dietary Supplement: Placebo
- Daidzein (Experimental): 10g soy protein isolated plus 50mg daidzein powder patch by mouth everyday for 6 months
  Interventions: Dietary Supplement: Daidzein
- Genistein (Experimental): 10g soy protein isolated plus 50mg genistein powder patch by mouth everyday for 6 months
  Interventions: Dietary Supplement: Genistein

INTERVENTIONS:
Dietary Supplement: Placebo — 10g soy protein isolated per day
  Arms: Placebo
Dietary Supplement: Daidzein — 50mg daidzein +10g soy protein isolated per day
  Arms: Daidzein
Dietary Supplement: Genistein — 50mg genistein +10g soy protein isolated per day
  Arms: Genistein

SUMMARY:
Many studies showed that soy foods or soy isoflavones can lower the risk of cardiovascular disease (CVD), osteoporosis and some cancers, but few human studies assessed effects of purified isoflavone components (genistein and daidzein) on glucose metabolism. This double-blinded, randomized, placebo-controlled trial will examine the effects of purified genistein and daidzein on glucose metabolism in prediabetic or diabetic women. One hundred and eighty eligible women age 30-70 years(without any treatment of diabetic drugs) will be recruited and randomly allocated into the following three arms: Placebo (10g isolated soy protein, ISP); Genistein (10g ISP + 50mg genistein); Daidzein (10g ISP + 50mg daidzein) per day for 6 mo. Fasting glucose, lipids, insulin, inflammation marks and post-load for glucose and insulin will be determined at 0, 3th, and 6th month. Changes in these indices will be compared among the three groups.

DETAILED DESCRIPTION:
Subjects were Chinese adult women, age 30-70 year, with an FG concentration ranging from 5.6 to 7.0 mmol/L or 2-h PG concentration ranging from 7.8-11.0 mmol/L or with newly diagnosed diabetes not requiring medication treatment according to a doctor's suggestion or participants did not willing to take medication themselves, and managed their diabetes just with a stable diet and exercise. Women were excluded if they had a history of coronary heart disease, stoke, thyroid disease, severe liver, lung, or gastrointestinal tract diseases; were currently or in the past 8 weeks used hypoglycemic or lipid-lowering or weight-reduction agents; were occurrence of diabetic complications; use of hormone replacement therapy; allergy to soy;were long-term antibiotics users.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women aged 30-70 y
* Fasting glucose >=5.6 mmol/l; post-load glucose >=7.8 mmol/l

Exclusion Criteria:

* Diabetes renal diseases
* Confirmed CVD, chronic liver,kidney diseases,Thyroid disease
* Medications affecting glucose or lipid metabolism

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan-bin Ye, MD, Principal Investigator — Sun Yat-sen University; Yu-ming Chen, PhD, Study Director — Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: the recruitment period last about half a year,and the types of location are clinic of endocrinology and nutritional clinic
Groups:
- Placebo: the placebo group were given 10g soy protein isolated without isoflavones
- Daidzein: Daidzein group were given 10g soy protein isolated and 50mg purify daidzein
- Genistein: Genistein group were given 10g soy protein isolated and 50mg purify genistein
Period: Overall Study
Arm/Group | Placebo | Daidzein | Genistein
Started | 54 | 55 | 56
Completed | 47 | 50 | 54
Not Completed | 7 | 5 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Other:Depression | 1 | 0 | 0
Not completed — Other: Colon cancer | 1 | 0 | 0
Not completed — Other: Stroke | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Daidzein | Genistein | Total
Number analyzed (Participants) | 54 | 55 | 56 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 43 | 42 | 128
  >=65 years | 11 | 12 | 14 | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 56.31 (11.07) | 56.36 (9.90) | 57.02 (9.68) | 56.57 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 56 | 165
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 54 | 55 | 56 | 165

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Fasting Plasma Glucose
Description: (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline,6 months
Population: the number of participants for analysis was determined by intention to treat
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Placebo Group: All participants were received 10g soy protein isolated without isoflavones daily
- Daidzein Group: All participants were received 10g soy protein isolated plus 50mg purify daidzein daily
- Geinstein Group: All participants were received 10g soy protein isolated plus 50mg purify genistein daily
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
percentage of change | -1.80 (13.5) | -1.00 (12.61) | -4.89 (11.79)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Null hypothesis: There are no difference in the difference of changes in plasma glucose. Power calculation: The sample size of 55 subjects per group provided about 90% power to detect a significant change in the FG concentration of 8 mg/dL (7%) by using a general assumption of a 2-tailed a level of 0.05 and allowing for a 20% withdrawal rate; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.7981, 95% CI 2-sided [-6.6569 to 5.0607], Standard Error of Mean 2.422
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 3.0842, 95% CI 2-sided [-2.7486 to 8.9171], Standard Error of Mean 2.411
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 3.8823, 95% CI 2-sided [-1.9234 to 9.6881], Standard Error of Mean 2.399

2. Primary Outcome: Percentage Change in 120-minutes Postload Plasma Glucose
Description: (6th month value-baseline value)/baseline*100%
Time Frame: Baseline, 6 months
Population: All participants were determinted by intention to treat
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
percentage of change | -4.90 (20.67) | -3.13 (20.60) | -5.59 (24.23)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -1.7696, 95% CI 2-sided [-11.9308 to 8.3916], Standard Error of Mean 4.2000
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 0.6929, 95% CI 2-sided [-9.4232 to 10.8091], Standard Error of Mean 4.1818
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 2.4626, 95% CI 2-sided [-7.6067 to 12.5318], Standard Error of Mean 4.1624

3. Primary Outcome: Percentage Change in HbA1C
Description: (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of participants analyzed was determinted by intention to treat.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
percentage of change | -1.38 (7.17) | -1.37 (5.99) | -1.30 (9.29)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.01174, 95% CI 2-sided [-3.5428 to 3.5194], Standard Error of Mean 1.45967
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -2.68659, 95% CI 2-sided [-6.2020 to 0.8288], Standard Error of Mean 1.45320
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -2.67485, 95% CI 2-sided [-6.174 to 0.8243], Standard Error of Mean 1.44646

4. Primary Outcome: Percentage Change in AUC of Glucose
Description: values were from 75g glucose oral glucose tolerance test and caculated as (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of patticipants was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
percentage of change | -6.23 (14.06) | -3.27 (16.98) | -5.24 (17.96)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -2.9661, 95% CI 2-sided [-10.5857 to 4.6535], Standard Error of Mean 3.14977
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Odds Ratio, log = -0.9972, 95% CI 2-sided [-8.5830 to 6.5886], Standard Error of Mean 3.13581
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Median Difference (Net) = 1.9689, 95% CI 2-sided [-5.5817 to 9.5195], Standard Error of Mean 3.12126

5. Primary Outcome: Percentage Change in Fasting Plasma Insulin
Description: (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of participants was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
percentage of change | 25.27 (114.23) | 21.41 (91.23) | 6.06 (78.26)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis; Mean Rank = 1.442

6. Primary Outcome: Percentage Change in HOMA-IR
Description: HOMA-IR was calculated with the homeostasis model assessment for insulin resistance,and it is caculated as the following equation: HOMA-IR=FIns×FG/22.5, where FIns represents fasting insulin in microunits per milliliter, and FG is in millimoles per liter. The percentage change was caculated as (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of participants for analysis was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
Percentage of change | 22.83 (107.41) | 21.60 (98.88) | -0.22 (64.03)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis; Mean Ranks = 1.895

7. Primary Outcome: Percentage Change in QUICKI
Description: QUICKI is the abbreviation of Quantitative Insulin Sensitivity Check Index,and it is a marker to evaluate insulin sensitivity in HOMA model.It is calculated by using the following equation: 1/(logFIns +logFG),where FIns represents fasting insulin in microunits per milliliter, and FG is in millimoles per liter.
  The percentage change was caculated as (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of participants for analysis was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
Percentage of change | 2.32 (19.47) | 0.18 (15.60) | 6.29 (17.77)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis; Mean Ranks = 2.169

8. Primary Outcome: Percentage Change in Total Cholesterol
Description: (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of participants for analysis was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
Percentage of change | 2.85 (40.06) | -0.59 (11.90) | -0.64 (15.83)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 3.4370, 95% CI 2-sided [-8.444 to 15.318], Standard Error of Mean 4.9113
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 3.4809, 95% CI 2-sided [-8.3475 to 15.3092], Standard Error of Mean 4.8896
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 0.0439, 95% CI 2-sided [-11.7296 to 11.8174], Standard Error of Mean 4.8669

9. Primary Outcome: Percentage Change in Triglyceride
Description: (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of participants for analysis was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
Percentage of change | 5.93 (45.50) | 3.43 (38.90) | -1.56 (39.15)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis; Mean ranks = 1.031

10. Primary Outcome: Percentage Change in High Density Lipoprotein Cholesterol
Description: (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
Percentage of change | 3.18 (20.40) | 1.36 (15.21) | 2.15 (14.54)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 1.8185, 95% CI 2-sided [-6.0057 to 9.6426], Standard Error of Mean 3.2343
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 1.0276, 95% CI 2-sided [-6.7619 to 8.8170], Standard Error of Mean 3.2199
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.7909, 95% CI 2-sided [-8.5442 to 6.9624], Standard Error of Mean 3.2050

11. Primary Outcome: Percentage Change in Low Density Lipoprotein Cholesterol
Description: (6th month value-baseline value)/baseline value*100%
Time Frame: Baseline, 6 months
Population: The number of participants for analysis was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 54 | 55 | 56
Percentage of change | 1.08 (24.46) | -0.93 (21.21) | 1.86 (19.39)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 2.0122, 95% CI 2-sided [-8.0721 to 12.0964], Standard Error of Mean 4.1686
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.7716, 95% CI 2-sided [-10.8111 to 9.2679], Standard Error of Mean 4.1501
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -2.7837, 95% CI 2-sided [-12.7767 to 7.2092], Standard Error of Mean 4.1309

12. Secondary Outcome: Total Urinary Isoflavones
Time Frame: 3 months
Population: The number of participants for analysis was determinted by the participants who provided the urine samples at the 3-month test.
Measure: Geometric Mean (Standard Deviation); unit: ug/ml
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 46 | 52 | 50
ug/ml | 8.538 (10.153) | 25.818 (31.780) | 15.467 (22.022)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.4437, 95% CI 2-sided [-0.6416 to -0.2458], Standard Error of Mean 0.1001
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.1986, 95% CI 2-sided [-0.3956 to -0.0016], Standard Error of Mean 0.09986
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 0.2451, 95% CI 2-sided [0.0544 to 0.4358], Standard Error of Mean 0.09648

13. Secondary Outcome: Urinary Daidzein
Description: Urinary daidzein excretion
Time Frame: 3 months
Population: The number of participants for analysis was determinted by the number of participants who provided urine samples at the 3-month test
Measure: Geometric Mean (Standard Deviation); unit: ug/ml
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 46 | 52 | 50
ug/ml | 3.34 (4.81) | 11.80 (11.14) | 3.73 (8.83)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.6353, 95% CI 2-sided [-0.8617 to -0.4089], Standard Error of Mean 0.1146
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Net) = 0.0282, 95% CI 2-sided [-0.2003 to 0.2568], Standard Error of Mean 0.1156
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 0.6635, 95% CI 2-sided [0.4419 to 0.8851], Standard Error of Mean 0.1121

14. Secondary Outcome: Urinary Genistein
Description: Urinary genistein excretion
Time Frame: 3 months
Population: The number of participants for analysis was determinted by the number of participants who supplied the urine samples at the 3-month test
Measure: Geometric Mean (Standard Deviation); unit: ug/ml
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 46 | 52 | 50
ug/ml | 1.32 (1.72) | 1.89 (2.59) | 6.54 (8.97)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.1557, 95% CI [-0.3911 to 0.0796], Standard Error of Mean 0.1190
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Net) = -0.6060, 95% CI 2-sided [-0.8414 to -0.3707], Standard Error of Mean 0.1190
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -0.4503, 95% CI 2-sided [-0.6804 to -0.2202], Standard Error of Mean 0.1163

15. Secondary Outcome: Total Energy Intake at Follow-up
Description: The energy intake was evaluated by 3 days dietary records.
Time Frame: an average of the 24 weeks follow-up period which were evalutated on baseline,12 week and 24 week.
Population: The number of participants for analysis was determinted by intention to treat
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Placebo Group | Daidzein Group | Geinstein Group
Number analyzed (Participants) | 47 | 50 | 54
kcal | 1575 (575) | 1473 (294) | 1579 (367)
Statistical Analysis 1: Comparison: Placebo Group vs Daidzein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 102.4, 95% CI 2-sided [-99.3 to 304.1], Standard Error of Mean 83.4
Statistical Analysis 2: Comparison: Placebo Group vs Geinstein Group; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Net) = -3.8, 95% CI 2-sided [-203.7 to 196.1], Standard Error of Mean 82.6
Statistical Analysis 3: Comparison: Daidzein Group vs Geinstein Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = -106.2, 95% CI 2-sided [-305.1 to 92.8], Standard Error of Mean 82.2

ADVERSE EVENTS:
Time Frame: We collected 10 cases of other adverse events which were mild to moderate in severity in the 6 months intervention period.
Arm/Group | Placebo | Daidzein | Genistein
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 4/54 | 4/55 | 2/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Daidzein (N=55) | Genistein (N=56)
vignal bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
hyperplasia of mammary glands (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
thirsty (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A relative long time of recruitment leading to a little different in dietary intakes among subjects;The menstrual period will leading to different estradiol;The different severity of the diabetes leading to the different dropout percentage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes